CLINICAL TRIAL: NCT04268836
Title: Vision Improvement for Patients With Age-Related Macular Degeneration
Acronym: AMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Optimal Acuity Corporation (Industry)
Collaborators: Bochner Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OAC #001
Record Dates: First submitted 2018-01-16; First posted 2020-02-13 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-04

CONDITIONS: Age-related Macular Degeneration
Keywords: dry AMD; wet AMD; neovascular AMD; age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, unmasked clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Patients will be treated by the Optimal Acuity Clear-K Low Vision Aid System.
  Interventions: Device: Optimal Acuity Clear-K® Low Vision Aid System treatment

INTERVENTIONS:
Device: Optimal Acuity Clear-K® Low Vision Aid System treatment — The treatment involves irradiation of the cornea with low energy light in a treatment pattern that produces corneal shape change.

SUMMARY:
The purpose of this study is to determine whether the Optimal Acuity Clear-K® Low Vision Aid System provides a safe and effective treatment to improve vision for patients with age-related macular degeneration.

DETAILED DESCRIPTION:
The Optimal Acuity Clear-K® Low Vision Aid System treats corneas with near infrared light in order to change the modulus of small volumes of anterior stromal corneal tissue. The change of modulus produces a change of corneal stiffness and shape that modifies the distribution of light onto the retina. Light rays are redirected from dysfunctional areas of the retina that have been damaged by age-related macular degeneration (AMD) to functional areas of the retina, thereby improving patient vision.

200 AMD patients meeting eligibility requirements will be treated. The study will record and analyze pre-treatment (Tx) and post-Tx examinations with follow-up extending to 24 months post-Tx. Analysis will include descriptive statistics and measures of correlation between outcomes and patient baseline characteristics.

The primary objective of the study is to evaluate the safety and effectiveness of Clear-K® treatment in providing vision improvement to AMD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Any race
3. Patient is at least 50 years old.
4. Patient has diagnosed dry or wet age-related macular degeneration in one or both eyes, as verified by a complete ocular examination by a retina specialist; the full ocular examination, including optical coherence tomography (OCT) measurements, should be part of the patient's file.
5. Wet AMD eyes should have an inactive disease state (i.e., there is no clinical or OCT evidence of wet AMD disease activity).
6. Patient is pseudophakic or is phakic with no clinically significant cataract in eye(s) to be treated..
7. Patient has manifest refraction, spherical equivalent (MRSE) between -1.50 D to 1.50 D in eye(s) to be treated.
8. Patient has moderate to severe vision impairment due to dry age-related macular degeneration with best spectacle-corrected distance visual acuity (CDVA) of 20/80 or worse (decimal = 0.25 or less; logMAR ≥ 0.60) in the better eye.
9. Patient has CDVA of 20/400 or better (decimal = 0.05 or greater; logMAR ≤ 1.30) in the worse eye.
10. Patient has normal corneal surface topography on videokeratography (i.e., without distorted or unclear corneal mires) in both eyes.
11. Patient is not a contact lens (CL) wearer.
12. Patient is willing and able to comply with all examinations.
13. Patient must be competent to sign an informed consent form before study entry.

Exclusion Criteria:

1. Corneal disease or disorder in either eye;
2. Corneal topographic astigmatism greater than 2.00 D (mean value within 3.0 mm optical zone);
3. Pathological retinal morphology in either eye that completely affects the entire 10° (3 mm diameter) of the retina centered on the foveola (as evaluated by optical coherence tomography);
4. Potential Visual Acuity (PVA) in both eyes that is not improved by at least three lines compared to CDVA;
5. Increased intraocular pressure (above 20 mm Hg), glaucoma or history of glaucoma; and
6. Presence or history of any other condition or finding that, in the opinion of the investigator, makes the patient unsuitable as a candidate for study participation or that may confound the outcome of the study.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-09 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Best spectacle-corrected distance visual acuity (CDVA) changes from baseline to 24 months post-Tx | Through study completion, an average of 2 years
  CDVA will be measured using ETDRS letter scoring both pre-Tx and post-Tx with follow-up to 24 months post-Tx

SECONDARY OUTCOMES:
Visual Function Questionnaire (VFQ)-25 quality of life assessment | Through study completion, an average of 2 years
  The VFQ-25 instrument will be used to assess patient quality of life measures.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Berry, PhD, Study Director — Optimal Acuity Corporation
Locations (1):
- 1929 Bayview Ave., Suite 117, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No